CLINICAL TRIAL: NCT03563989
Title: STENTYS Xposition S in the Treatment of Chronic Total Artery Occlusion (SXS-CTO)
Brief Title: STENTYS Xposition S in the Treatment of Chronic Total Artery Occlusion
Acronym: SXS-CTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K171009J
Record Dates: First submitted 2018-05-28; First posted 2018-06-20 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-05

CONDITIONS: Chronic Total Occlusion; Coronary Artery Disease
Keywords: Chronic total occlusion; Self-expandable stent; Percutaneous coronary intervention; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stentys Xposition S Self-Apposing stent (Experimental): STENTYS Xposition S Sirolimus Eluting Self-Apposing Coronary Stent System
  Interventions: Device: Implantation of Stent (PCI)
- Conventional Balloon-expandable stent (Active Comparator): Conventional Balloon-expandable drug eluting stents in effect at the time of the study, in compliance with applicable contracts made between Hospital and suppliers.
  Interventions: Device: Implantation of Stent (PCI)

INTERVENTIONS:
Device: Implantation of Stent (PCI) — Treatment of CTO with Percutaneous Coronary Intervention (PCI) Patients are randomized to receive either self-expandable stent or balloon expandable stent

SUMMARY:
Intro: Chronic total occlusions (CTO) are the most severe coronary lesions. Negative distal vessel remodeling occurs in these lesions, leading to reduction of artery diameter. Treatment of CTO with percutaneous coronary intervention (PCI) is associated with good clinical outcomes. However, QCA and IVUS studies showed a notable lumen and vessel enlargement distal to recanalized CTO. In addition, optical tomography (OCT) studies showed high rates of stent strut malapposition and incomplete stent strut coverage after CTO PCI. The Stentys Xposition S is a self-apposing stent device which lowers stent strut malapposition rates. Its safety and effectiveness has been demonstrated in STEMI and stable coronary patients but never investigated in CTO lesions.

Hypothesis/Objective To investigate whether self-expanding stents are more effective than balloon-expandable stents for reducing stent malapposition at 6 months after implantation in patients with CTO undergoing percutaneous coronary intervention.

Method Pilot randomized study. Patients are randomized to receive either self-expandable stent or balloon expandable stent to perform CTO-PCI. Follow-up coronary angiography is performed at 6 months post-PCI. Stent malapposition is evaluated by OCT.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* CTO referred for PCI
* Diameter of the Target vessel for PCI between 2.5 and 4.5mm
* Agreement to participate and signed informed consent after information
* Affiliation to Social Security System
* French comprehension

Exclusion Criteria:

* Pregnant women, breast-feeding,
* History of an allergic reaction or significant sensitivity to any stent component or to contrast dye
* Intrastent CTO
* Major calcifications in the CTO
* Inclusion in another interventional study
* Person under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
strut malapposition at six months measured by OCT | 6 months after CTO-PCI

SECONDARY OUTCOMES:
percentage of uncovered struts | 6 months after CTO-PCI
lumen diameter (mm) | 6 months after CTO-PCI
Restenosis | 6 months after CTO-PCI
Angina pectoris | 6 months after CTO-PCI
Dyspnea | 6 months after CTO-PCI
Mortality | 6 months after CTO-PCI
Stroke | 6 months after CTO-PCI
Stent thrombosis | 6 months after CTO-PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION